CLINICAL TRIAL: NCT06847178
Title: A Trial Investigating the Efficacy and Safety of LC-Z300-01 in Adults With Type 2 Diabetes
Brief Title: Efficacy and Safety of LC-Z300-01 in Chinese With Type 2 Diabetes
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: LC-Z300-01
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Diabetes; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Masks

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The total duration of the trial for individuals participating in this clinical trial is up to 30 weeks, including:
  1. 3-week screening period,
  2. 1-week run-in period (may be extended to a maximum of 8 weeks),
  3. 12-week double-blind randomized, controlled intervention period,
  4. 12-week switching to high-dose conversion, open-label intervention period,
  5. 2-week follow-up period. For subjects with an extended run-in period, the trial duration can be up to 37 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- low-dose LC-Z300-01 (Experimental): Experimental: placebo for runing-in + LC-Z300-01 Subjects will receive 12-weeks of low-dose LC-Z300-01 randamizedly and then 12 weeks of high-dose LC-Z300-01 in open-label.
  Interventions: Drug: Low-dose LC-Z300-01 twice daily in blinding; Drug: High-dose LCZ300-1 twice daily in open-label
- high-dose LC-Z300-01 (Experimental): Experimental: placebo for runing-in + LC-Z300-01 Subjects will receive 24-weeks of high-dose LC-Z300-01.
  Interventions: Drug: High-dose LC-Z300-01 twice daily in blinding; Drug: High-dose LCZ300-1 twice daily in open-label
- Placebo (Placebo Comparator): Experimental: placebo + LC-Z300-01 Subjects will receive 12-weeks of placebo radamizedly and then 12 weeks of high-dose LC-Z300-01 in open-label.
  Interventions: Dietary Supplement: Placebo twice daily in blinding; Drug: High-dose LCZ300-1 twice daily in open-label

INTERVENTIONS:
Dietary Supplement: Placebo twice daily in blinding — Administered placebo twice-daily for 12 weeks in blinding
  Other Names: Double-blind phase （placebo）
  Arms: Placebo
Drug: Low-dose LC-Z300-01 twice daily in blinding — Administered twice-daily for 12 weeks in blinding
  Other Names: Double-blind phase （LC-Z300-01）
  Arms: low-dose LC-Z300-01
Drug: High-dose LC-Z300-01 twice daily in blinding — Administered twice-daily for 12 weeks in blinding
  Other Names: Double-blind phase （LC-Z300-01）
  Arms: high-dose LC-Z300-01
Drug: High-dose LCZ300-1 twice daily in open-label — Administered high-dose LCZ300-1 twice-daily for 12 weeks in open-label
  Other Names: Open-label phase (LC-Z300-01)

SUMMARY:
This trial is conducted in China. The aim of the trial is to investigate the efficacy and safety of an Bamboo cane polysaccharide (oral LC-Z300-01) in subjects with type 2 diabetes.

DETAILED DESCRIPTION:
This trial is conducted in China. The aim of the trial is to investigate the efficacy and safety of an Bamboo cane polysaccharide (oral LC-Z300-01) in subjects with type 2 diabetes.

Considering the rights and interests, the trial is divided into two phases. The first phase is a double-blind group, in which subjects are randomly assigned to the blank control group, the low-dose experimental group, and the high-dose experimental group to observe the changes in glycosylated hemoglobin and CGMS compared with the baseline, as well as safety events.

The second phase is an open-label group, in which the three groups are willing to freely enter the high-dose experimental group and further observe recovery and safety.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age reach and over 18 years at the time of signing informed consent,
* Body mass index (BMI) between 18.0 and 35.0 kg/m^2 (both inclusive),
* Type 2 diabetes mellitus (as diagnosed clinically) before screening.
* hemoglobin A1c of 7.5 - 9.0% (both inclusive) as assessed by central laboratory on the day of screening,
* Treated with stable doses of oral antidiabetic drugs (OADs) , insulin or glucagon-like peptide-1 (GLP-1) receptor agonists (exenatide, liraglutide, etc.) within 3 months prior to screening;

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using a highly effective contraceptive method,
* Anticipated initiation or change in concomitant medication (for more than 14 consecutive days) known to affect weight or glucose metabolism (e.g. treatment with orlistat, thyroid hormones, or systemic corticosteroids),
* Any episodes (as declared by the participant or in the medical records) of diabetic ketoacidosis within 90 days before screening,
* Presence or history of pancreatitis (acute or chronic) within 180 days before screening,
* Any of the following: Myocardial infarction, stroke, hospitalization for unstable angina pectoris or transient ischaemic attack within 180 days before screening.

Chronic heart failure classified as being in New York Heart Association Class IV at screening,

* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within the past 90 days before screening or in the period between screening and randomisation. Pharmacological pupil dilation is a requirement unless using a digital fundus photography camera specified for non dilated examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events | From baseline week 0 to week 26
  The differences in adverse events between the patients taking the drug and the placebo group were observed during the double-blind and open-label phases.
Change in glycated haemoglobin (HbA1c) | From baseline week 0 to week 12 and to week 24
  During the double-blind and open-label phases, the changes in dynamic blood glucose and CGMS values of patients taking the medication compared with the baseline were observed and compared with those in the placebo group.

SECONDARY OUTCOMES:
Change in Time in Range (TIR) | From baseline week 0 to week 12 and to week 24
  During the double-blind and open-label phases, the changes in dynamic blood glucose and CGMS values of patients taking the medication compared with the baseline were observed and compared with those in the placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-fen Xie, Prof., Study Director — Shanghai Changzheng Hospital
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No